CLINICAL TRIAL: NCT02658344
Title: Multicenter, Randomized, Double-Blind, Placebo Controlled Phase Ⅱb Clinical Trial to Evaluate Efficacy and Safety of JOINTSTEM in Patients With Degenerative Arthritis
Brief Title: Clinical Trial to Evaluate Efficacy and Safety of JOINTSTEM in Patients With Degenerative Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: R-Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Jointstem2b
Record Dates: First submitted 2015-08-03; First posted 2016-01-18 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Degenerative Arthritis; Knee Osteoarthritis
Keywords: Stem cell; adipose tissue derived mesenchymal stem cell; osteoarthritis; degenerative arthritis; biostar; Rbio
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Jointstem (Experimental): Autologous Adipose Tissue derived MSCs
  Interventions: Biological: JOINTSTEM
- Saline solution (Placebo Comparator): Sodium chloride
  Interventions: Drug: Saline solution

INTERVENTIONS:
Biological: JOINTSTEM — Jointstem (Autologous Adipose Tissue derived MSCs 1x10^8cells/3ml), 1 time injection
  Other Names: Autologous Adipose Tissue derived MSCs 1x10^8cells/3ml
  Arms: Jointstem
Drug: Saline solution — Saline solution (Sodium chloride 9mg/ml), 1 time injection
  Other Names: Sodium chloride 9mg/ml
  Arms: Saline solution

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of autologous transplantation of Adipose Tissue derived Mesenchymal stem cells (MSCs) in patient with Knee Osteoarthritis.

DETAILED DESCRIPTION:
JOINTSTEM is an OA treatment that uses autologous adipose-derived mesenchymal stem cells. As it does not use allogenic tissues and is incubated without additional genetic modification or mechanical and chemical modification through differentiation, it is classified as 'autologous cell therapy' and is completely free of immunologic rejection.

It primarily aims to improve pain and joint function, and secondary, to regenerate cartilage. The intra-articular injection of JOINTSTEM is expected to stimulate the regeneration and growth of cartilage, and to innovatively improve pain and joint function with cartilage regeneration within six months.

The subjects of this therapy were regenerative patients with K&L grade 2~4 aged 18 or older. JOINTSTEM is expected to be used in patients who have significantly damage cartilage due to its cartilage regeneration ability, in addition to its improvement of pain and joint performance. A;sp. Patients who had already undergone knee arthroplasty can delay their additional surgery with the use of JOINTSTEM. For dose who still have their own cartilage, arthroplasty is not an immediate treatment option, and osteoporosis patients who cannot undergo arthroplasty due to their advanced age can receive JOINTSTEM.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older, male and female
2. Patients must consent in writing to participate in the study by signing and dating an informed consent document
3. Diagnosis of osteoarthritis by ACR osteoarthritis of the knee
4. Diagnosis of osteoarthritis by radiographic criteria of Kellgren and Lawrence grade 2-4
5. More than Grade 4 (0~10 point numeric scale) pain at least for 12 weeks
6. Diagnosis of osteoarthritis of class Ⅰ~Ⅲ by ACR(American College of Rheumatology Criteria) Global functional criteria
7. Patient who agree with contraception

Exclusion Criteria:

1. Preparing for Pregnancy or Pregnant women or lactating mothers.
2. Patients with Body Mass Index (BMI) > 35.
3. Patients with other disease including

   : Septic arthritis, Rheumatoid or Inflammatory joint disease, Crystalline disease (gout or pseudogout), Paget disease, Articular fractures, Ochronosis, Acromegaly, Hemochromatosis, Wilson's disease, Osteochondromatosis, Hereditary disorder
4. Patients with serious condition internal medicine disease
5. Patients with positive human immunodeficiency (HIV), hepatitis B (HBV), hepatitis C (HCV), syphilis at screening indicative of current of pass infection.
6. Patient with behavioral disorders, cognitive disorders and chronic mental symptoms
7. Patient with significant neurologic or psychiatric disorders
8. Patients who alcohol, drug abuse history
9. Patients who had participated in other clinical trials within 12 weeks prior to this study.
10. Patients who received any drug by intra-articular injection for treatment within 2 months prior to this enrollment.
11. Patients who experienced as the knee joint cartilage and stem cell therapy
12. Patients who the principal investigator considers inappropriate for the clinical trial due to any other reasons than those listed above
13. Patients who penicillin hypersensitivity reactions -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-07; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
WOMAC score | 24 weeks
  Pain, stiffness, and physical function of the knee will be measured by the Western Ontario and McMaster Universities (WOMAC)

SECONDARY OUTCOMES:
WOMAC 3 subscale | 24 weeks
  Pain, stiffness, and physical function of the knee will be measured by the Western Ontario and McMaster Universities (WOMAC)
KOOS (Knee Injury & Osteoarthritis Outcome Score) | 24 weeks
  Symptoms, pain and functionality of the knee joint will be evaluated via the Knee Injury and Osteoarthritis Outcome Score (KOOS)
SF(Short Form)-36 Score | 24 weeks
  The SF(Short Form)-36 Health Survey is a 36-item, patient-reported survey of patient health.
Global assessment of disease activity | 24 weeks
  Change From Baseline in Patient's & Physician's Global Assessment of Disease Activity Score at 12,24 weeks by 100mm VAS(Visual Analogue Scale)
Overall satisfaction | 24 weeks
  Patient's overall satisfaction on a 0-100mm VAS(Visual Analogue Scale)
X-ray | 24 weeks
  X-ray perform to measure with Kellgren-Lawrence grade
MRI scan | 24 weeks
  MRI perform to measure cartilage defect size change from baseline up to 24weeks
Arthroscopy evaluation | 24 weeks
  Arthroscopy performs to evaluate any change in cartilage defect at the time of cell injection, and at 24 weeks after injection
Histological evaluation | 24 weeks
  Biopsy specimens subject to safranin-O staining and immunohistochemistry for type I and II collagen. Thickness of the articular cartilage before and after injection measure, and specimens evaluate with ICRS(International Cartilage Repair Society) II by a blind histopathologist.
VAS | 24 weeks
  Pain of the knee will be measured by the 100mm Visual Analogue Scale (VAS)
IKDC | 24 weeks
  Symptoms, sports activities, and function of the knee will be measured by the International Knee Documentation Committee (IKDC)
ROM | 24 weeks
  change from baseline in knee flexion Range of Motion(ROM) at 12,24 weeks by physical examination
Quadriceps power | 24 weeks
  Change from baseline in quadriceps power at 12,24 weeks by physical examination
effusion | 24 weeks
  Change from baseline in 4-grade knee effusion at 12,24 weeks
Crepitus | 24 weeks
  Change from baseline in asymptomatic and symptomatic crepitus at 12,24 weeks by physical examination
Ligament laxity | 24 weeks
  Change from baseline in ligament laxity at 12,24 weeks by physical examination
Medial joint line tenderness | 24 weeks
  Change from baseline in 4-grade(none, mild, moderate, severe) medial joint line tenderness at 12,24 weeks by physical examination
Pes tenderness | 24 weeks
  Change from baseline in 4-grade(none, mild, moderate, severe) Pes tenderness at 12,24 weeks by physical examination

CONTACTS AND LOCATIONS:
Overall Officials: KANGIL KIM, M.D., Ph.D, Principal Investigator — KyungHee University Gangdong Hospital
Locations (2):
- South Korea (2):
  - KyungHee University Gangdong Hospital, Seoul
  - GangNam Severance Hospital, Seoul

REFERENCES:
- [Result] Lee WS, Kim HJ, Kim KI, Kim GB, Jin W. Intra-Articular Injection of Autologous Adipose Tissue-Derived Mesenchymal Stem Cells for the Treatment of Knee Osteoarthritis: A Phase IIb, Randomized, Placebo-Controlled Clinical Trial. Stem Cells Transl Med. 2019 Jun;8(6):504-511. doi: 10.1002/sctm.18-0122. Epub 2019 Mar 5. PMID 30835956